CLINICAL TRIAL: NCT05309317
Title: The Effect of Virtual Simulation Game on Improving Nursing Students' Knowledge and Skills Regarding Prevention of Catheter- Associated Urinary Tract Infection
Brief Title: Preventing Catheter-Associated Urinary Tract Infections With a Virtual Simulation Game
Acronym: CAUTI-VSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Mercan Annak, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 57440
Record Dates: First submitted 2022-03-09; First posted 2022-04-04 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Catheter-Associated Urinary Tract Infection; Nurse's Role
Keywords: Virtual Simulation Game; Catheter-Associated Urinary Tract Infection; Nursing Education; Nursing Students

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAUTI-VSG (Experimental): Preventing Catheter-Associated Urinary Tract Infections with a Virtual Simulation Game
  Interventions: Other: Virtual Simulation Game for the Prevention of Catheter-Associated Urinary Tract Infections; Other: Ongoing education
- Control group (Active Comparator): Training on "CAUTI Prevention"
  Interventions: Other: Ongoing education

INTERVENTIONS:
Other: Virtual Simulation Game for the Prevention of Catheter-Associated Urinary Tract Infections — A training on "Prevention of CAUTI" will be held for the experimental and control groups. The experimental group will be able to play a seven-day virtual simulation game devised by the researcher to prevent CAUTI.
  Arms: CAUTI-VSG
Other: Ongoing education — Only a course on "Prevention of CAUTI" will be given to the control group.

SUMMARY:
Objective: The purpose of this study was to investigate the effectiveness of a virtual simulation game in improving nursing students' knowledge and abilities in preventing catheter-associated urinary tract infection (CAUTI).

Method: The study was designed as a parallel-group, randomized controlled trial. A pre-test on knowledge and abilities will be administered to all students participating in the study. Following the pre-test evaluation, a training session on "CAUTI Prevention" will be held. The present training approach (lecture method) in the curriculum will be employed in this session. Following the training, the students in the sample group will be randomly divided into the experimental group (students using virtual simulation game application) and the control group (students learning with the existing education method) based on their general weighted grade averages using the stratified randomized approach. The experimental group will play the virtual simulation game for seven days. Knowledge and competence assessments (post-test) of the control and experimental groups will be conducted seven days following the training. The virtual simulation game application will be evaluated by the students in the experimental group after the post-test evaluations. The students' positive, negative, and constructive feedback on the virtual simulation game will be solicited during the assessment. In addition, these students will score in a 5-point Likert type to evaluate the statements about the virtual simulation game.

Hypothesis: H0-1: There is no difference in knowledge about preventing CAUTI between students using the virtual simulation game method and students in the control group.

H1-1: There is a difference in knowledge about preventing CAUTI between students using the virtual simulation game method and students in the control group.

H0-2: There is no difference in CAUTI prevention skills between students using the virtual simulation game method and students in the control group.

H1-2: There is a difference in CAUTI prevention skills between students using the virtual simulation game method and students in the control group.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in Nursing Profession Courses Practice-II for the first time
* To agree to participate in the study
* To have internet access and smartphone or computer

Exclusion Criteria:

* Not filling in the data collection forms of the research at any stage
* Answering the data collection forms of the research incomplete
* Not having received the first or last skill assessments
* Not attending the training on preventing CAUTI
* Not playing/completing the virtual simulation game

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-05-21 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Knowledge Level | Change from students' knowledge levels at seven days
  The investigator developed the "Knowledge Test on Preventing Catheter-Associated Urinary Tract Infection." There are 25 multiple-choice questions with five options on the test. The response to each question in the knowledge test will be scored out of 100 points, with 4 points being awarded for each correct answer. The overall score is based on a scale of 0 to 100. Higher scores imply that the student has a higher degree of knowledge.
Skill level | Change from students' skill levels at seven days
  The investigator developed the "Skills Assessment Checklist for Preventing Catheter-Associated Urinary Tract Infection." Emptying the collecting bag, mobilization, specimen collection, and removal of the urine catheter of the patient are the parts of the competency evaluation checklist. The stages on the skill evaluation checklist will be scored as "Applied" (3 points), "Partly Applied (Incorrect)" (2 points), "Partly Applied (Missing)" (2 points), and "Not Applied" (3 points) (1 point). The collecting bag emptying checklist has 13 steps (minimum 13, maximum 39 points), the mobilization checklist has 8 steps (minimum 8, maximum 24 points), the specimen collection checklist has 22 steps (minimum 22, maximum 66 points), and the urinary catheter removal checklist has 13 steps (minimum 22, maximum 66 points) (minimum 13, maximum 39 points). Higher scores imply that the student's skill level is improving.

SECONDARY OUTCOMES:
Opinions of the experimental group about the virtual simulation game | within 1 week after intervention
  The Virtual Simulation Game Application Evaluation Form is divided into two sections. Three open-ended questions regarding the virtual simulation game are asked in the first section (What are your positive thoughts about the virtual simulation game?, What are your negative thoughts about the virtual simulation game?, What are your suggestions about the virtual simulation game?) The Virtual Simulation Game Technology Acceptance Questionnaire (SSO-TKA) is included in the second section, and it was created using the Technology Acceptance Model as a guide. The SSO-TKA contains 21 items that are used to assess the game's ease of use (applicability-15 items) and perceived utility (usability-6 items). Students will use a 5-point Likert scale to rate the items relevant to the virtual simulation game (1: Strongly disagree, 2: Disagree, 3: Undecided, 4: Agree, 5: Strongly Agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No